CLINICAL TRIAL: NCT02804841
Title: D-activating Decline- Exploring the Effects of Vitamin D3 Supplementation on Cognitive Function in Community Dwelling Healthy Older Adults- A Pilot Study
Brief Title: Effects of Vitamin D3 Supplementation on Cognitive Function in Community Dwelling Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Dublin, Trinity College (Other)
Responsible Party: Principal Investigator, Maria O'Sullivan, Associate Professor, University of Dublin, Trinity College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: UniDublinTC
Record Dates: First submitted 2016-05-20; First posted 2016-06-17 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-11

CONDITIONS: Healthy
Keywords: Vitamin D supplementation; Cognitive function; Physical function; Successful ageing; Prevention; Cholecalciferol; Dementia; Muscle mass
MeSH Terms: conditions — Dementia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Healthy, Community Dwelling; Aged 60-80 years; Cholecalciferol -Vitamin D3, 4000 international units (IU) on alternating days.
  Interventions: Dietary Supplement: Cholecalciferol -Vitamin D3
- Placebo (Placebo Comparator): Healthy, Community Dwelling; Aged 60-80 years; Placebo -gel capsule containing no vitamin D on alternating days.
  Interventions: Other: Placebo -gel capsule containing no vitamin D.

INTERVENTIONS:
Dietary Supplement: Cholecalciferol -Vitamin D3
  Arms: Intervention
Other: Placebo -gel capsule containing no vitamin D.
  Arms: Placebo

SUMMARY:
Ireland is predicted to have the highest older adult population growth of any European Union country. A substantial economic and social challenge of this projected growth is the increased incidence of cognitive impairment and the likelihood of progression to dementia. Dementia's, such as Alzheimer's disease, typically have a long prodromal stage with brain changes identifiable from the earliest stages of neuropathology, providing an opportunity for intervention. Switching to a strategy of earlier identification and prevention would significantly reduce prevalence and the associated cost.

The purpose of this pilot study is to evaluate the use of vitamin D supplements in community dwelling older adults as a lifestyle approach that may support cognitive and physical functioning. The research will incorporate several stages including an initial in-depth screening process, a novel and sensitive cognitive battery, 6 month double blind placebo controlled intervention of vitamin D3 (cholecalciferol) and a concluding participant feedback interview.

These results will be used to assess the feasibility of recruiting and assessing community dwelling older adults for extensive nutrition related cognitive studies.

ELIGIBILITY:
Inclusion Criteria:

* Community Dwelling healthy volunteers
* Ability to provide written consent.

Exclusion Criteria:

* Measures low or high serum vitamin D, defined as < 15nmol/L or >125nmol/L
* Current use of supplemental vitamin D ≥800 international units/d
* Screen positive for cognitive impairment using the Telephone Cognitive Screen (TCogS)
* Measured hypercalcaemia, defined as corrected serum calcium > 2.7nmol/l
* Hyperparathyroidism
* Epilepsy
* Stroke
* Renal disease
* Schizophrenia
* Bipolar affective disorder
* Recurrent psychotic depression
* Alcohol and drug abuse within the past 5 years
* Anti-convulsants
* Anti-psychotic medications
* Significant hearing difficulties even when wearing hearing aid
* Illness that caused permanent decrease in memory or other mental function

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-11; Primary Completion 2016-05 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Global Cognitive Function | 26 weeks
  Global cognitive function will be assessed using the validated Montreal Cognitive Assessment for all participants
Executive Function | 26 weeks
  Executive function will be assessed according to the validated Trails Making Task Part A and B
Memory | 26 weeks
  Episodic memory will be assessed according to the Wescher Memory Scale
Attention and Visual Reasoning | 26 weeks
  Attention and visual memory will be assessed using 2 validated measures: the Sustained Attention to Response Task and the Cambridge Mental Disorders of the Elderly Examination Visual Reasoning Test

SECONDARY OUTCOMES:
Muscle strength | 26 weeks
  Muscle strength in the participants will be assessed using a clinical dynamometer to measure grip strength
Physical function | 26 weeks
  Physical function will be assessed using the Timed up and Go measure
Systemic inflammation | 26 weeks
  Serum will be analysed for levels of specific cytokines
Change in Blood Level of Vitamin D (25-hydroxyvitamin D) | 0, 12 and 26 weeks
  Serum will be analysed for change in levels from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Maria O'Sullivan, PhD, Principal Investigator — The University of Dublin, Trinity College; Brian Lawlor, MD, Principal Investigator — The University of Dublin, Trinity College
Locations (1):
- University of Dublin, Trinity College, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No